CLINICAL TRIAL: NCT04413812
Title: Fostering Exercise After Bariatric Surgery
Acronym: FREEBASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lia Bally (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Professor, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FREEBASE
Record Dates: First submitted 2020-04-16; First posted 2020-06-04 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Bariatric Surgery; Physical Activity
Keywords: Training Intervention; Health Competence; Active Lifestyle; Bariatric Surgery; Lifestyle Modification
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized single-centre open-label clinical trial with two parallel groups. The randomization will be stratified according to age, sex, current BMI, surgical procedure, and educational level using a dedicated software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will participate in a 3-months training programme focusing on health competence related outcomes.
  Interventions: Behavioral: FREEBASE exercise programme
- Control Group (No Intervention): The control group does not participate in the exercise programme but undergoes identical outcome assessments.

INTERVENTIONS:
Behavioral: FREEBASE exercise programme — The exercise programme will be initialized 1-10 months following bariatric surgery and last for 3 months. The programme will be mainly delivered in two groups consisting of 10-12 subjects each and will be held in the facilities of a fitness studio and remotely at home. The programme consists of 24 units (two per week, the lesson in the fitness studio lasting for 75 minutes and the remote lesson lasting for 45 minutes.This is due to the COVID-19-related social distancing restrictions. The intervention combines the following elements: a) exercise training in a group, b) interactive workshops on basic knowledge of training sciences and techniques of behavior change and c) an individual exercise counselling session.
  The programme will be medically supervised and the content will be taught and instructed by members of the research team qualified in exercise science and sports physiology.
  Arms: Experimental Group

SUMMARY:
While the benefits of engagement in regular physical activity after bariatric surgery has been established in various studies, little is known about the effectiveness of an interdisciplinary intervention including nutritional and psychological advice, hands-on training experience and motivational education to promote long-term adherence to a self-motivated active lifestyle in the bariatric surgery population.

This randomized pilot intervention study called Fostering Exercise After Bariatric Surgery (FREEBASE) explores the efficacy of an interdisciplinary approach to promote physical activity-related health competence and an active lifestyle after bariatric surgery.

DETAILED DESCRIPTION:
Bariatric surgery is quickly emerging as a standard treatment for people with obesity stage II and III (BMI ≥35 kg/m2) because of its beneficial long-term effects on body weight and obesity-related comorbidities. In Switzerland, approximately 5,000 bariatric surgeries are performed every year. There is a growing body of evidence demonstrating that engagement in physical activity benefits the bariatric surgery population in many aspects. These entail the prevention of surgery-induced metabolic complications such as sarcopenia and osteopenia on the one hand, but also the mitigation against the commonly observed weight regain and relapse of metabolic comorbidities. Despite these obvious health benefits, inactivity and poor health literacy are common problems amongst people who underwent bariatric surgery. Although the Swiss healthcare system offers well designed post-operative follow-up programmes, exercise is currently not to being considered. Additionally the lower educational level of bariatric surgery patients is a well known problem. Addressing physical activity-related health competence and self-empowerment in this population currently remains an unmet need.

Previous studies investigating exercise interventions in the bariatric surgery population have demonstrated efficacy on metabolic outcomes but also indicated that adherence wanes over time. To overcome the challenge of changing lifestyle in a sustainable way, individuals need to have a complex set of abilities, skills, knowledge, motivation and willingness. In Germany, diverse models have been developed to describe this specific set of competences, all inspired by the concept of health literacy, which is internationally recognised in research and clinical practice.

Physical activity-related health competence comprises three components: (1) Movement competence, enabling individuals to meet the movement-related requirements of physical activities (e.g. motor abilities, motor skills for cycling or gymnastics) (2) control competence for physical activity enabling people to gear their own activity to achieve positive effects in health and well-being, and (3) physical activity-specific self-regulation competence enabling individuals to be regularly active, which involves both motivational and volitional factors. The relevance of physical activity-related health competence for the promotion of an active lifestyle has been demonstrated in various studies in healthy and physical inactive adults at metabolic risk. However, the concept has not yet been addressed in the bariatric surgery population. The investigators therefore hypothesize, that targeting the various components of physical activity-related health competence by means of a comprehensive exercise programme has the potential to result in a more effective promotion of physical activity in the bariatric surgery population, thereby benefitting their long-term health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Bariatric surgery within the past 1-6 months according to the guidelines of the Swiss Society for the Study of Morbid Obesity and Metabolic Disorders (SMOB)
* Willingness to comply with study-related activities
* Literate in German

Exclusion Criteria:

* Incapacity to give informed consent
* Contraindication to participation in the study exercise programme as judged by the clinical investigator or treating physical
* Physical or physiological condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the clinical investigator or treating physical
* Evidence of malnutrition as judged by the clinical investigator or treating physician
* Pregnancy, planned pregnancy, or breast feeding (females of childbearing potential are advice to use safe-contraception for up to 18 months post-bariatric surgery as part of usual care)
* Illicit or prescription drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical activity-related health competence. | The questionnaires will be completed at baseline, after completion of the exercise program (visit 2, at 10-12 weeks) and at the follow-up (visit 3, at 16-18 weeks).
  The physical activity-related health competence will be assessed using items from different areas (self-efficacy, self-control, emotional attitudes, cognitive attitudes, motivational competence, control of physical load, affect regulation). A composite score will be calculated as the mean score of the individual areas. For each area, the mean score of its items assessed on a 5-point Likert scale ranging from 1 (does not apply at all) to 5 (does apply exactly) will be calculated.

SECONDARY OUTCOMES:
Relative change from baseline in physical activity level. | Physical activity will be measured during one week at baseline and during one week at follow-up (visit 3, at 16-18 weeks).
  Physical activity level will be assessed using accelerometry and is defined as the overall daily mean acceleration (mg).
Change from baseline in self-reported physical activity. | The questionnaires will be completed at baseline, after completion of the exercise program (visit 2, at 10-12 weeks) and at the follow-up (visit 3, at 16-18 weeks).
  Self-reported physical activity will be assessed using the German Physical Activity, Exercise, and Sport Questionnaire "Bewegungs- und Sportaktivität Fragebogen; BSA-F". This questionnaire asks for frequency and duration of daily physical activities such as walking, cycling, garden work, house work, caring for others in the last four weeks. The frequency and duration for each question are multiplied and the products are added up in an overall physical activity index (in minutes/week).
Change from baseline in self-reported sport and exercise activity. | The questionnaires will be completed at baseline, after completion of the exercise program (visit 2, at 10-12 weeks) and at the follow-up (visit 3, at 16-18 weeks).
  Self-reported sport and exercise activity will be assessed using the German Physical Activity, Exercise, and Sport Questionnaire "Bewegungs- und Sportaktivität Fragebogen; BSA-F". This questionnaire includes questions about regular exercise and sport activities. People can indicate up to three exercise and sport activities and indicate frequency and duration in the last four weeks. The frequency and duration for the named exercise and sport activity are multiplied and the products are added up to an exercise and sport activity index (in minutes/week).
Absolute change in 6-min walking distance (m) | The test will be conducted at baseline and at visit 2 (after 10-12 weeks).
Absolute change in Time (s) in the "Timed up and go" test. | The test will be conducted at baseline and at visit 2 (after 10-12 weeks).
Absolute change in Time (s) in the "Unilateral hip bridge" test | The test will be conducted at baseline and at visit 2 (after 10-12 weeks).

OTHER OUTCOMES:
Change from baseline in health status | The questionnaires will be completed at baseline, after completion of the exercise program (visit 2, at 10-12 weeks) and at the follow-up (visit 3, at 16-18 weeks).
  The health status will be assessed using the German questionnaire for health status assessment "Allgemeiner Gesundheitszustand"
Change from baseline in vitality. | The questionnaires will be completed at baseline, after completion of the exercise program (visit 2, at 10-12 weeks) and at the follow-up (visit 3, at 16-18 weeks).
  Vitality will be assessed using the German questionnaire "Vitalitätsskala" ("subjective vitality scale") on a 7-point Likert scale ranging vom 1 (not applicable at all) to 7 (very applicable).
Change from baseline in self-concordance. | The questionnaires will be completed at baseline, after completion of the exercise program (visit 2, at 10-12 weeks) and at the follow-up (visit 3, at 16-18 weeks).
  The self-concordance will be assessed on a 6-point Likert scale ranging from 1 (does not apply at all) to 6 (applies exactly).
Change from baseline in the intention to perform physical activity. | The questionnaires will be completed at baseline, after completion of the exercise program (visit 2, at 10-12 weeks) and at the follow-up (visit 3, at 16-18 weeks).
  The intention to perform physical activity will be assessed on a 10-point Likert scale ranging from 1 (I have no such intention) to 10 (I have this intention very strongly).
Participant satisfaction. | Within the first week after completion of the exercise program.
  The satisfaction will be assessed using a self-designed feedback questionnaire. The overall satisfaction is assessed on a 5-point Likert scale ranging from 1 (not satisfied at all) to 5 (very satisfied).
Perception of usefulness of the program. | Within the first week after completion of the exercise program.
  The usefulness will be assessed on a 5-point Likert scale ranging from 1 (not useful at all) to 5 (very useful).
Change from baseline in self-regulation competence. | The questionnaire will be completed at baseline, after completion of the exercise program (at 10-12 weeks) and at follow-up (at 16-18 weeks).
  The self-regulation competence will be calculated as the mean score of the items "self-efficacy", "self-control", "emotional attitudes", "cognitive attitudes", and "motivational competence". Each item is assessed on a 5-point Likert scale ranging from 1 (does not apply at all) to 5 (applies exactly).
Change from baseline in control competence | The questionnaire will be completed at baseline, after completion of the exercise program (visit 2, at 10-12 weeks) and at follow-up (visit 3, at 16-18 weeks).
  The control competence will be calculated as a mean score of the items "control of physical load" and "affect regulation". Each item is assessed on a 5-point Likert scale ranging from 1 (does not apply at all) to 5 (applies exactly).

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD, PhD, Principal Investigator — University Hospital Bern & University of Bern, Bern, Switzerland
Locations (1):
- Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No